CLINICAL TRIAL: NCT00360802
Title: The Effectiveness of Cognitive Behavioral Treatment and Mindfulness Based Stress Reduction for Chronic Low Back Pain Treated in Pain Clinics
Brief Title: Effectiveness of Cognitive Behavioral Treatment and Mindfulness Based Stress Reduction (MBSR) for Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kovacs Foundation (Other)
Collaborators: Spanish Back Pain Research Network (REIDE) (Other); Fondo de Investigacion Sanitaria (Other); Universitat Autonoma de Barcelona (Other)
Responsible Party: Jenny Moix, Professor, Universidad Autónoma de Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: FK-FIS-22
Record Dates: First submitted 2006-08-04; First posted 2006-08-07 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2009-05

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; cognitive-behavioral therapy; Mindful Based Stress Reduction; pain clinics; anxiety; quality of life; chronic pain
MeSH Terms: conditions — Anxiety Disorders; Chronic Pain | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- CBT (Active Comparator): Cognitive Behavioral Treatment
  Interventions: Behavioral: Cognitive Behavioral Treatment
- MBSR (Active Comparator): Mindfulness Based Stress Reduction
  Interventions: Behavioral: Mindfulness Based Stress Reduction

INTERVENTIONS:
Behavioral: Cognitive Behavioral Treatment — Behavioral treatment to reduce pain in chronic back pain patients
  Arms: CBT
Behavioral: Mindfulness Based Stress Reduction — Behavioral treatment to reduce pain in chronic back pain patients
  Arms: MBSR

SUMMARY:
The primary purpose of this study is to determine the effectiveness of two psychological techniques in chronic low back pain patients treated in hospital pain clinics. The techniques are: cognitive behavioral treatment and mindfulness based stress reduction (MBSR). This is a multiple site project in which patients come from 16 different pain clinics throughout Spain. The control group is formed by patients under usual medical treatment at pain clinics. The two intervention groups also receive usual medical treatment at pain clinics plus one psychological therapy treatment. The sample size is 330 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain and failed back surgery patients
* With or without referred or radiated pain
* Who are between 18 and 70 years of age (inclusive)

Exclusion Criteria:

* Patients with red flags for systemic disease or criteria for surgery
* With intolerable intensity of pain despite 6 weeks or more of non-surgical treatment
* With pain that appears only on walking and disappears with sitting, persists after 6 months of conservative treatment, and is a possible spinal stenosis
* Under psychological or psychiatric treatment
* Unable to fill out the questionnaires
* Have received cognitive behavioral treatment in the past
* Have ongoing work litigation or are in the process of obtaining permanent disability.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Degree of improvement in: anxiety, quality of life | immediately after therapy, at 3 months, and at 12 months

SECONDARY OUTCOMES:
Degree of improvement in: pain, disability, catastrophizing, depression, anger, analgesic medication, satisfaction with treatment received | immediately after therapy, at 3 months, and at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M. Kovacs, MD, PhD, Study Chair — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Jenny Moix, PhD, Principal Investigator — Departamento de Psicología Básica, Universidad Autónoma de Barcelona, Bellaterra, Barcelona 08193, Spain; María José Martín, Study Director — Hospital Mutua de Terrasa, Terrasa 08221, Spain; María Angeles Pastor, Study Director — Hospital General y Universitario de Alicante, Alicante 03010, Spain; María Isabel Casado, PhD, Study Director — Hospital 12 de Octubre, Madrid 28041, Soain; Carlos Peña, PhD, Study Director — Hospital Universitario Marqués de Valdecilla, Santander 39008, Spain; Andrés Martín, BS, Study Director — Hospital de Son Llatzer, Palma de Mallorca 07198, Spain; Gema Rodríguez, Study Director — Hospital Severo Ochoa, Leganés, Madrid 28911, Spain; Francisco Javier Cano, PhD, Study Director — Hospital Universitario Virgen del Rocío, Sevilla 41013, Spain; Milena Gobbo, BS, Study Director — Fundación Hospital Alcorcón, Madrid 28922, Spain; Almudena Mateos, BS, Study Director — Fundación Hospital Alcorcón, Madrid 28922, Spain; Carla Casals, BS, Study Director — Hospital de Figueres, Figueres 17600, Spain
Locations (1):
- Universidad Autónoma de Barcelona, Dept. Psicología Básica, Evolutiva y de la Educación, Bellaterra, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Deyo RA, Weinstein JN. Low back pain. N Engl J Med. 2001 Feb 1;344(5):363-70. doi: 10.1056/NEJM200102013440508. No abstract available. PMID 11172169
- [Background] van Tulder MW, Ostelo R, Vlaeyen JW, Linton SJ, Morley SJ, Assendelft WJ. Behavioral treatment for chronic low back pain: a systematic review within the framework of the Cochrane Back Review Group. Spine (Phila Pa 1976). 2000 Oct 15;25(20):2688-99. doi: 10.1097/00007632-200010150-00024. PMID 11034658
- [Background] Basler HD, Jakle C, Kroner-Herwig B. Incorporation of cognitive-behavioral treatment into the medical care of chronic low back patients: a controlled randomized study in German pain treatment centers. Patient Educ Couns. 1997 Jun;31(2):113-24. doi: 10.1016/s0738-3991(97)00996-8. PMID 9216352
- [Derived] Moix J, Kovacs FM, Martin A, Plana MN, Royuela A; Spanish Back Pain Research Network. Catastrophizing, state anxiety, anger, and depressive symptoms do not correlate with disability when variations of trait anxiety are taken into account. a study of chronic low back pain patients treated in Spanish pain units [NCT00360802]. Pain Med. 2011 Jul;12(7):1008-17. doi: 10.1111/j.1526-4637.2011.01155.x. Epub 2011 Jun 13. PMID 21668743
- See also: Spanish Back Pain Research Network site that describes objectives and projects of its members — http://www.reide.org